CLINICAL TRIAL: NCT01905293
Title: Individual Differences in Children's Susceptibility to Overeating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: R03DK091492 (NIH)
Record Dates: First submitted 2013-07-11; First posted 2013-07-23 (Estimated); Last update posted 2013-07-23 (Estimated); Status verified 2013-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 100% portion size (Experimental): 100% portion size condition
  Interventions: Other: Feeding Study
- 150% portion size (Experimental): 150% portion size condition
  Interventions: Other: Feeding Study
- 200% portion size (Experimental): 200% portion size condition
  Interventions: Other: Feeding Study

INTERVENTIONS:
Other: Feeding Study

SUMMARY:
The portion size of foods has been identified as an important determinant of energy intake in children. It remains to be determined to what extent child weight status and the relative reinforcing value of food may interact with the obesogenic food environment to affect energy intake. The primary aim of this study was to compare energy intake at a meal in normal-weight and obese children when the portion size of palatable, energy-dense foods and a sugar-sweetened beverage was systematically increased. We hypothesized that increasing the portion size of all foods and the beverage at a meal will lead to a significant increase in energy intake in both normal-weight and obese children. Obese children, however, will show a significantly greater increase in energy intake than will normal-weight children. A second aim of this study was to test if children's response to increases in portion size was affected by how reinforcing they find food to be. We hypothesized that, when controlling for BMI, children who find food very reinforcing relative to nonfood alternatives will show a significantly greater increase in energy intake than will children who find food less reinforcing.

DETAILED DESCRIPTION:
The prevalence of childhood and adolescent obesity has reached an all-time high. There is a pressing need to better understand the behavioral mechanisms that control appetite and eating in children and to identify children who are most susceptible to overeating in the current obesogenic food environment. Obesogenic environments offer convenient access to large portions of palatable, energy-dense foods. The portion size of foods has been identified as an important determinant of energy intake in adults and children. While portion size effects have been found in heterogenous groups of healthy individuals, some evidence points to possible individual differences in the magnitude of children's responsiveness to large food portions. For example, data from a previous laboratory study suggest that overweight and obese children may be particularly vulnerable to overeating when presented with large food portions. Further, the magnitude of a portion size effect on intake may also depend on how reinforcing (or rewarding) children find food to be. It is possible that the relative reinforcing value of food may interact with environmental cues, such as the portion size of food, to affect children's energy intake when large portions of palatable, energy-dense foods are available. The primary aim of this study is to compare the effects of increasing the portion size of all foods and a beverage served at a meal on energy intake in normal-weight and obese children. A second aim is to test if children who find food very reinforcing relative to an appealing nonfood alternative will show a significantly greater increase in energy intake in response to increasing portion sizes than will children who find food less reinforcing. The findings from this study are expected to extend previous findings to test how environmental factors, such as food portion size, may interact with individual differences in weight status or food reinforcement to affect energy intake in children.

ELIGIBILITY:
Inclusion Criteria:

* 8 to 10 years of age
* normal-weight or obese
* like most foods that were served in the study

Exclusion Criteria:

* serious medical conditions or medication use known to affect appetite, food intake, and body weight
* developmental or psychiatric conditions
* learning disability
* sight or hearing impairment
* food allergies or nutrient intolerances (including lactose intolerance)

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2011-05; Primary Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Total energy intake | Up to 3 weeks

SECONDARY OUTCOMES:
Energy intake from food | Up to 3 weeks
Energy intake from beverage | Up to 3 weeks
Percent estimated energy requirement (%EER) | Up to 3 weeks
Relative reinforcing value of food (RRVF) | Up to 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tanja VE Kral, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: National Institute of Diabetes and Digestive and Kidney Diseases — http://www2.niddk.nih.gov